CLINICAL TRIAL: NCT03372486
Title: Effect of Ultra-low Dose Naloxone During Supraclavicular Brachial Plexus Block on the Anti-nociceptive Criteria of Post-operative Opioid in Orthopedic Upper Limb Surgeries
Brief Title: Effect of Ultra-low Dose Naloxone During Supraclavicular Brachial Plexus Block on Post-operative Opioi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD ∕ 17.07.95
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Upper Extremity Trauma
MeSH Terms: interventions — Bupivacaine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine plus naloxone (Active Comparator): Patients will receive brachial plexus block using bupivacaine plus naloxone.
  Interventions: Drug: Bupivacaine plus naloxone
- Bupivacaine (Placebo Comparator): Patients will receive brachial plexus block using bupivacaine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine plus naloxone — Patients received 20 mL bupivacaine 0.5% plus 100 ng naloxone (1ml) in 2ml saline.(naloxone ampoule 0.4mg will dilute in 400ml of saline then 1ml of it will dilute in 10 ml saline, so each ml will have 100ng naloxone)
  Arms: Bupivacaine plus naloxone
Drug: Bupivacaine — Patients will be injected ultrasound guided in their brachial plexus by 20 mL bupivacaine 0.5% plus 3 ml of saline
  Arms: Bupivacaine

SUMMARY:
Effective post-operative pain control can reduce patient morbidity and affect the patient outcome. Brachial plexus block is one of them, a popular and widely employed regional nerve block technique for perioperative anesthesia and analgesia for surgery of the upper extremity.

Different drugs have been used as adjuvants with local anesthetics in brachial plexus block to achieve quick, dense and prolonged block like Morphine, Pethidine, Clonidine, Dexmedetomidine.

Naloxone is opioid antagonists which could selectively block the excitatory effects of opioids. it release endorphins and also displace endorphins from receptor site .it also reduce the opioid induced side effects, such as vomiting, nausea, pruritus, and respiratory depression.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of ultra-low dose of naloxone when added to bupivacaine %.05 in supraclavicular brachial plexus block in orthopedic upper limb surgery and if it enhances the anti-nociceptive effect of post-operative opioid

Effect of naloxone on anti-nociceptive criteria of post -operative opioid will be estimated by detecting the interval between each analgesic dose of post-operative opioid.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical state class Ι and II
* Elective upper limb orthopedic surgery (hand, forearm and elbow)
* Duration of surgery ≤180 min
* BMI ≤30 kg/m2

Exclusion Criteria:

* History of allergy to the drug of the study.
* Coagulation disorders
* Infection at the puncture site.
* Pregnancy
* Opioid abuse.
* Abuse of tranquilizers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Effect of ultra-low dose naloxone on the post operative opioid | for 48 hours after surgery
  by estimate the analgesic requirements of opioids and the interval between each opioid dose in 48 hour post operative

SECONDARY OUTCOMES:
Duration of sensory block | For 48 hours after surgery
  will be defined as the time interval between the complete sensory block (complete absence of pinprick response) and first experience with postoperative pain
Duration of motor block | For 48 hours after surgery
  defined as the time interval between complete paralysis (Lovett rating scale = 0) and complete recovery (Lovett rating scale = 6)
Onset time of sensory block | For 48 hours after surgery
  defined as the time between the end of the last injection and complete absence of pinprick response in all nerve distribution
Onset time of motor block | For 48 hours after surgery
  defined as the time between the end of the last injection and complete paralysis (Lovett rating scale = 0) in all nerve distributions
Severity of post-operative pain | For 48 hours after surgery
  will be measured by visual analogue scale (VAS) where 0 was equal to no pain and 10 indicated the worst possible pain
1st time of analgesic request | For 48 hours after surgery
  First need for rescue opioid after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Doaa G Diab, MD, Principal Investigator — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Central Hospital, emergency Unit, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided